CLINICAL TRIAL: NCT00449163
Title: Phase II Study of Avastin, Irinotecan, High Dose 24 Hour Continuous Intravenous Infusion of Floxuridine and Leucovorin in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy and Bevacizumab in Treating Patients With Stage IV Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by University of Miami Institutional Review Board
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060042; SCCC-2005145 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20060252 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Floxuridine; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Chemotherapy and Bevacizumab (Experimental): Treatment cycle is 6 weeks, 2 weeks of consecutive treatment followed by 1 week of rest and 2 weeks of treatment followed by one week of rest. Treatment will be administered weekly, 4 out 6 weeks, on days 1, 8, 22 and 29:
  * Bevacizumab: 7.5mg/kg via intravenous (IV) infusion on Days 1 and 22;
  * Irinotecan: 110 mg/m^2 via IV infusion on Days 1, 8, 22, 29;
  * Leucovorin: 500 mg/m^2 via IV infusion on Days 1, 8, 22 and 29;
  * Floxuridine: 120 mg/kg over continuous infusion on Days 1, 8, 22 and 29.
  Interventions: Biological: Bevacizumab; Drug: Floxuridine; Drug: Irinotecan; Drug: Leucovorin

INTERVENTIONS:
Biological: Bevacizumab
  Other Names: Avastin
Drug: Floxuridine
  Other Names: 5-fluorodeoxyuridine
Drug: Irinotecan
  Other Names: Irinotecan Hydrochloride; Camptosar
Drug: Leucovorin
  Other Names: Leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, floxuridine, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with bevacizumab works in treating patients with stage IV colorectal cancer.

DETAILED DESCRIPTION:
For the purpose of this study treatment cycle consist of six weeks, 2 weeks of consecutive treatment followed by 1 week of rest and 2 weeks of treatment followed by one week of rest. Treatment will be administered weekly, 4 out 6 weeks, on days 1, 8, 22 and 29 according to the schedule. There will be no treatment delivered on weeks 3 & 6 (Days 15 and 36).

Disease will be evaluated by CT scan at the completion of every two cycles. Patients with complete response (CR), or partial response (PR), will be evaluated for possible surgical resection. Patients who become operable will continue to be evaluated for survival and disease relapse. Patients with stable disease (SD), and those with less than pCR after surgery should continue chemotherapy until radiographic evidence of tumor progression is identified or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have stage IV, histologically confirmed diagnosis of Adenocarcinoma of the colon.
2. Patients must have bi-dimensionally measurable disease since the purpose of this study is to determine efficacy of treatment.
3. Patients must be previously untreated.
4. Patients must be over the age of 18 years.
5. Patients may not be pregnant. Patients of childbearing years must be using contraception.
6. Patients must have ECOG performance status of 0-1 or KPS of at least 70.
7. Patients must have life expectancy of ≥ two months.
8. Patients must have a white blood cell count of ≥1000/mm³ ANC > 1.0, platelets > 100,000/mm³.
9. Patients must have adequate renal function as documented by a serum creatinine of ≤ 1.5 mg/dl.
10. Patients must have a bilirubin of ≤ 1.5 mg/dl and an SGOT of ≤ three times normal for patients with no liver disease, and ≤ five times normal for those with liver metastases.
11. Patients must be informed of the investigational nature of the study and give written informed consent.
12. Patients must have indwelling central venous catheter or good peripheral intravenous catheter, preferably a port-a-cath.
13. Patients may have had prior surgery for their colorectal cancer. Patients must be at least 8 weeks beyond surgery and recovered from all effects of surgery.
14. Patients enrolled in this study may have a history of prior malignancy (5 years ago) provided that the patient is currently disease-free.

Exclusion Criteria:

1. Patients who have had prior chemotherapy or radiation therapy for their colorectal cancer, with exception of adjuvant chemo/radiation therapy.
2. Patients receiving concomitant radiation, hormonal therapy, chemotherapy, or immunotherapy.
3. Patients receiving any investigational drug within 30 days prior to start of this study.
4. Patients with serious underlying medical illnesses (including Congestive Heart Failure New York Heart Association Functional Classification 2-4) or active infection.
5. Patients with central nervous system metastasis must have completed radiation prior to entry into this protocol.
6. Patients with psychiatric conditions or associated conditions which would make participating in this study dangerous to their health.
7. Patients with uncontrolled hypertension.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bach Ardalan, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Result] Phase II study of bevacizumab (B), camptosar (I), high-dose 24-hour continuous intravenous infusion of floxuridine (F) and leucovorin (L) in patients with previously untreated metastatic colon cancer. (B-IFL) B. Ardalan, M. Feagans, D. Mezentsev, C. Jones, P. R. Subbarayan, G. Walker, M. Sapp, K. Stephenson, J. Ness, D. Franceschi, and A. Livingstone Journal of Clinical Oncology 2009 27:15S, e15114-e15114

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 25 subjects were enrolled however; data were analyzed for only 22 of the subjects enrolled.
Period: Overall Study
Arm/Group | Combination Chemotherapy and Bevacizumab
Started | 25
Completed | 22
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Combination Chemotherapy and Bevacizumab
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival up to 2 Years
Description: Percentage of patients with overall survival times of up to 2 years
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Chemotherapy and Bevacizumab
Number analyzed (Participants) | 22
percentage of participants | 61 [27 to 83]

2. Secondary Outcome: Response Rate (Complete Response and Partial Response)
Description: Percentage of patients achieving complete response or partial response per RECIST criteria ver 1.0
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Chemotherapy and Bevacizumab
Number analyzed (Participants) | 21
percentage of participants | 67 [43 to 85]

3. Secondary Outcome: Median Progression-free Survival in Months
Description: Median number of months subjects achieved progression-free survival
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Chemotherapy and Bevacizumab
Number analyzed (Participants) | 21
months | 13 [8.4 to 15]

4. Secondary Outcome: Rate of Toxicity in Study Participants
Description: Evaluation the safety and toxicities of protocol regimen as evidenced by the rate of serious adverse events in study participants.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Combination Chemotherapy and Bevacizumab
Number analyzed (Participants) | 22
percentage of participants | 50

ADVERSE EVENTS:
Description: Only serious adverse events (Grade 3 and 4) reported.
Arm/Group | Combination Chemotherapy and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 5/22
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Chemotherapy and Bevacizumab (N=22)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 4
Diarrhea (Gastrointestinal disorders) | 3 — Grade 3
Fatigue (General disorders) | 2 — Grade 3
Port Site Thrombosis (Surgical and medical procedures) | 2 — Grade 3
Small Bowel Obstruction (Gastrointestinal disorders) | 2 — Grade 3
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 — Grade 3
DVT (Vascular disorders) | 3 — Grade 3
Infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
A total of 25 subjects were enrolled however; data were analyzed for 22 subjects only. Study was terminated early by the University of Miami Institutional Review Board.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes